CLINICAL TRIAL: NCT01268020
Title: An Exploratory, Open-label, Non-randomized Phase 0 Study to Evaluate [18F]-FMH3 by Positron Emission Tomography (PET) for Quantization of the Receptor Histamine-3 in Human
Brief Title: Evaluation of [18F] FMH3 and PET as a Marker of Histamine-3 Receptor Activity in Subjects With AD Compared w/ HC
Acronym: FMH3
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Institute for Neurodegenerative Disorders (Other)
Responsible Party: Principal Investigator, Danna Jennings, MD, Principal Investigator, Institute for Neurodegenerative Disorders
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: FMH3-01
Record Dates: First submitted 2010-12-28; First posted 2010-12-29 (Estimated); Last update posted 2013-11-11 (Estimated); Status verified 2013-11

CONDITIONS: Alzheimer Disease
Keywords: Alzheimer; AD
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- [18F]-FMH3-01 PET Imaging (Experimental): Subjects will be injected with up to 5 mCi and not to exceed 5.5mCi (not >10% of 5 mCi limit) or 2 ug of [18F]-FMH3, whichever is greatest.
  Interventions: Drug: [18F]-FMH3

INTERVENTIONS:
Drug: [18F]-FMH3 — Subjects will be injected with up to 5 mCi and not to exceed 5.5mCi (not >10% of 5 mCi limit) or 2 ug of [18F]-FMH3, whichever is greatest.

SUMMARY:
The underlying goal of this study is to assess [18F]-FMH3 PET imaging as a tool to evaluate the activity of the H3 receptor in the brain of Alzheimer Disease (AD) research participants

DETAILED DESCRIPTION:
Approximately 10 subjects with Alzheimer disease (AD) and 8 healthy control (HC)subjects will be recruited to participate in this study. All subjects will undergo written informed consent and a screening evaluation including baseline clinical laboratory testing, a baseline physical and neurological evaluation and baseline cognitive evaluations. Subjects will be asked to undergo a bolus injection of [18F]-FMH3. Subjects will undergo serial PET imaging scans and plasma sampling for measurement of [18F]-FMH3 in plasma (both protein bound and free) over a period of up to 8 hours. The primary imaging outcome measure will be the brain regional distribution volumes expressed as a brain tissue to plasma ratio of the radioligand, [18F]-FMH3.

At least 2 weeks following the initial imaging visit, subjects may be asked to return for a second injection and scanning procedure to evaluate the reproducibility of the imaging measure using this procedure. Subjects may decline to participate in the second scan.

ELIGIBILITY:
Inclusion Criteria:

The following criteria will be met for inclusion of AD subjects in this study:

* The participant is 50 years or older.
* Written informed consent is obtained.
* Participants have a clinical diagnosis of probable Alzheimer disease in accordance with the DSM-IV-TR and according to (NINCDS/ADRDA) criteria.
* Clinical Dementia Rating Scale score ≤ 2.
* Modified Hachinski Ischemia Scale score of ≤ 4.
* Geriatric Depression Scale (GDS) ≤ 10.
* For females, non-child bearing potential or a negative urine or blood pregnancy test on day of [18F]-FMH3 injection.

The following criteria will be met for inclusion of healthy control subjects in this study:

* The participant is 18 years or older.
* Written informed consent is obtained.
* Negative history of neurological or psychiatric illness based on evaluation by a research physician.
* Clinical Dementia Rating score = 0.
* For females, non-child bearing potential a negative urine or blood pregnancy test on day of [18F]-FMH3 injection.

Exclusion Criteria:

Alzheimer's subjects will be excluded from participation for the following reasons:

* The subject has a clinically significant abnormal laboratory value and/or clinically significant unstable medical or psychiatric illness
* The subject has any disorder that may interfere with drug absorption, distribution, metabolism, or excretion.
* The subject has evidence of clinically significant gastrointestinal, cardiovascular, hepatic, renal, hematological, neoplastic, endocrine, neurological, immunodeficiency, pulmonary, or other disorder or disease.

Healthy control subjects will be excluded from participation for the following reasons:

* The subject has a clinically significant abnormal laboratory value and/or clinically significant unstable medical or psychiatric illness.
* The subject has evidence of clinically significant gastrointestinal, cardiovascular, hepatic, renal, hematological, neoplastic, endocrine, neurological, immunodeficiency, pulmonary, or other disorder or disease.
* The subject has any disorder that may interfere with drug absorption, distribution, metabolism, or excretion.
* The subject has any contraindication to MRI examination, e.g. metal implants or phobia as determined by the onsite radiologist performing the scan.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2010-12; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
To assess the dynamic uptake and washout of 18F-FMH3 | 1 year
  To assess the dynamic uptake and washout of [18F]-FMH3, an imaging marker targeting the histamine H3 receptor in brain, using positron emission tomography (PET) in subjects with Alzheimer (AD) and healthy controls (HC).

CONTACTS AND LOCATIONS:
Overall Officials: Danna Jennings, MD, Principal Investigator — Institute for Neurodegenerative Disorders
Locations (1):
- Institute for Neurodegenerative Disorders, New Haven, Connecticut, United States